CLINICAL TRIAL: NCT06938555
Title: The RolE of Prolonged Nightly faSTing to Improve Sleep and cOgnition in bREast Cancer Survivors (RESTORE)
Brief Title: The RolE of Prolonged Nightly faSTing to Improve Sleep and cOgnition in bREast Cancer Survivors
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dorothy Sears, Executive Director and Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00021379
Record Dates: First submitted 2025-03-28; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Survivor; Cancer Related Cognitive Difficulties; Sleep; Quality of Life
Keywords: breast cancer; breast cancer survivor; brain fog; prolonged nightly fasting; nationwide; remote; non-invasive; health education; sleep; quality of life
MeSH Terms: conditions — Breast Neoplasms; Mental Fatigue; Health Education

STUDY DESIGN:
Intervention Model Description: One group will be assigned to Prolonged Nightly Fasting (PNF) and Health Education videos, the other group will be assigned to Health Education videos.
Who Masked: Investigator
Masking Description: Statistician will also be masked to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolonged Nightly Fasting and Health Education Videos (Experimental): Participants in the Prolonge + HED condition will receive both the Prolonged Nightly Fasting and the Health Education Video interventions.
  Interventions: Behavioral: Prolonged Nightly Fasting; Behavioral: Health Education Videos
- Health Education Videos Only (Active Comparator): Participants in the Health Education Only condition will participate in only the Health Education Video intervention. Investigators will provide materials about Prolonged Nightly Fasting to these participants at the end of the study.
  Interventions: Behavioral: Health Education Videos

INTERVENTIONS:
Behavioral: Prolonged Nightly Fasting — At the start of the intervention (week 1) PNF participants will be asked to engage in fasting (14 hours a night, starting no later than 8pm) six nights a week (for the 8-week study duration). Participants will be asked to track their fasting start/stop times on a tracking sheet provided by study staff. During the nightly fast, participants will be allowed to drink water, coffee or tea (without dairy or sweeteners). Study staff will meet with participants via phone for weekly check-in calls (~10-15 mins) to collect weekly fasting start/stop dates/times (entered into REDCap); alternately, participants may elect to email or text their fasting start/stop date/times to the study staff.
  Arms: Prolonged Nightly Fasting and Health Education Videos
Behavioral: Health Education Videos — Provision of HED is a retention strategy and can influence outcomes. Thus, all participants will receive HED. Each week, participants will receive hyperlinks to videos focused on health educational content unrelated to fasting, diet and outcome measures. Participants will be asked to view the videos (~10-15 min) prior to their weekly check-in calls with the study staff (~5-10 mins for HED-Only Control group). They will receive each week's videos on a Monday, and receive a reminder to view on Friday. Study staff will follow a scripted HED weekly check-in call to ensure consistency of data collected. Weekly topics are as follows: W1: Internet safety, W2: Sun safety, W3: Home safety, W4: Driving safety, W5: Hydration, W6: Dental health, W7: Working environment, W8: Communication. Data collected on electronic forms during all participant/staff check-in calls will be stored in participant-specific ASU Dropbox files.

SUMMARY:
The investigators are interested in finding out how Prolonged Nightly Fasting (PNF) and/or health education may impact health and cancer recovery for breast cancer patients and survivors.

DETAILED DESCRIPTION:
The purpose of this innovative, remotely-delivered pilot randomized controlled trial (RCT) is to explore the use of an 8-week prolonged nightly fasting (PNF) intervention, as compared to a Health Education-Only (HED-Only) control condition, among ethnically and racially diverse (≥50% Black, Hispanic, and/or Native American) breast cancer survivors (BCSs) with cancer-related cognitive impairment (CRCI) to examine changes in cognitive function, sleep, insomnia and health-related quality of life (i.e., mental and physical). Additionally, intervention feasibility will be assessed among the PNF participants. All participants will receive health education (HED) throughout. BCSs living with CRCI (N=60) will be recruited nationwide and randomized 1:1 into the PNF or HED-Only groups. Linear mixed models will be used to compare outcome changes in the PNF group compared to HED-Only group (Aims 1-3); descriptive and qualitative analyses will be used in the Exploratory Aim.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. diagnosed with breast cancer (all stages included)
3. ≥3 months post neoadjuvant or adjuvant chemotherapy (maintenance or palliative systemic therapy is included)
4. score ≤30 or lower on the Patient Reported Outcome Measurement Information System Cognitive Function Short Form 8a (sr-CRCI)
5. able to speak/understand English
6. have access to a computer and Wi-Fi
7. live within the United States
8. Identifies as female
9. willing and able to fully participate in the study

Exclusion Criteria:

1. type 1 diabetes
2. actively enrolled in formal diet/weight loss program
3. previous bariatric surgery
4. eating disorder history
5. night shift work
6. pregnant, breast feeding, or trying to get pregnant
7. dementia, psychological, psychiatric, or neurological diagnoses
8. active brain or central nervous system disease
9. prior or current use of memory enhancing medications
10. history or current brain radiation
11. frequently fasting for 12+ hours every night

13) history of hypoglycemia 14) depression screening on PHQ9 with a score of 20 or greater across all 9 questions OR anything other than 0 on question 9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must identify as women
Enrollment: 60 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Examine PNF-induced changes in cognitive function as compared to the HED-Only control condition. | Baseline (T1) and 8-week end point (T2) data collection
  The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) will be used to assess subjective cognitive function using a scale of 0-156
Examine PNF-induced changes in cognitive function as compared to the HED-Only control condition. | Baseline (T1) and 8-week end point (T2) data collection
  The Montreal Cognitive Assessment (T-MoCA) will be used to assess objective cognitive assessment using a scale of 0-22

SECONDARY OUTCOMES:
Examine PNF-induced changes in sleep (i.e., duration, quality) and insomnia as compared to the HED-Only Control condition. | Baseline (T1) and 8-week end point (T2) data collection
  Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep using a scale of 0-21
Examine PNF-induced changes in sleep (i.e., duration, quality) and insomnia as compared to the HED-Only Control condition. | Baseline (T1) and 8-week end point (T2) data collection
  Insomnia Severity Index (ISI) will be used to assess insomnia using a scale of 0-28
Examine PNF-induced changes in quality of life as compared to the HED-Only Control condition. | Baseline (T1) and 8-week end point (T2) data collection.
  Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS Global-10) questionnaire will be used to measure health-related quality of life (i.e., mental health, physical health). It uses a scale of 0-20.

OTHER OUTCOMES:
Exploratory Aim: Explore acceptability of the PNF intervention | 8-week end point (T2) data collection
  participant adherence to protocol
Exploratory Aim: Explore acceptability of the PNF intervention | 8-week end point (T2) data collection
  participant retention
Exploratory Aim: Explore acceptability of the PNF intervention | 8-week end point (T2) data collection
  qualitative interviews
Covariate Measure: eating behaviors | Baseline (T1) and 8-week end point (T2) data collection.
  Rapid Eating Assessment for Participants -- Shortened Version (REAPS) will be used to assess food intake quantity and quality changes. This uses a scale of 13-39

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Sears, PhD, Principal Investigator — Arizona State University; Sarah James, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Protocol and consent state, "De-identified data collected as a part of this study will not be shared with other investigators or industry partners for future research purposes."
  This is a pilot study and only aggregated data may be shared.